CLINICAL TRIAL: NCT01786642
Title: Assessment of the Efficacy of Tracheal Oxygen Administration During Bronchoscopy - a Phase II Trial.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Marc Decramer, MD, PhD, KU Leuven
Other Study IDs: AETOB
Record Dates: First submitted 2013-02-01; First posted 2013-02-08 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Hypoxaemia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- conscious: bronchoscopy without sedative drugs
- conscious sedation: bronchoscopy under midazolam

SUMMARY:
The aim of the present study is to measure the time to correction of O2 saturation when in case of desaturation below 90%, O2 administration is switched from the nasal to the tracheal route at a similar flow rate.

DETAILED DESCRIPTION:
The development of a flexible bronchoscope with a channel dedicated to O2 administration might allow optimization of the oxygen supplementation during bronchoscopy, which reduces the risk of per- and peri-procedural hypoxemia. The investigators will conduct a pilot study corroborating the hypothesis that tracheal supplementation of oxygen during flexible bronchoscopy is advantageous in comparison to nasal cannula supplementation.

The concept of our trial consists of a mono-centric observational study performed in the endoscopy suite of the Respiratory Division, University Hospitals Leuven. All patients will be given informed consent before inclusion.

The aim of the present study is to measure the time to correction of O2 saturation when in case of desaturation below 90%, O2 administration is switched from the nasal to the tracheal route at a similar flow rate.

ELIGIBILITY:
Inclusion Criteria:

* patients referred for flexible bronchoscopy

Exclusion Criteria:

* broncho-alveolar lavage
* endobronchial plugging

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients referred for flexible bronchoscopy
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-12 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Time to correction of SpO2 | procedure

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Dooms, Md PhD, Study Director — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University hospitals leuven, Leuven, Belgium